CLINICAL TRIAL: NCT01566474
Title: Melatonin Associated to Acid Inhibition for Chemoprevention in Barret Esophagus: a Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aragon Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICS10/0273
Record Dates: First submitted 2012-03-28; First posted 2012-03-29 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Omeprazole; Melatonin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin + omeprazole (Experimental): Omeprazole 40 mg/day + Circadin 6 mg/12 hours. Patients will take the Omeprazole capsule once in the morning before breakfast together with 3 tables of 2 mgs of Circadin (melatonin). In the evening, before dinner, patients will take 3 tablets of 2 mg of Circadin.
  Interventions: Drug: Melatonin
- omeprazole (Active Comparator): Omeprazole 40 mg/day alone. Patients will take the capsule once in the morning before breakfast. This is the standard therapy for patients suffering from Barrett's esophagus.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Omeprazole 40 mg/day alone. Patients will take the capsule once in the morning before breakfast. This is the standard therapy for patients suffering from Barrett's esophagus.
  Other Names: Generic omeprazole
  Arms: omeprazole
Drug: Melatonin — Omeprazole 40 mg/day + Circadin 6 mg/12 hours. Patients will take the Omeprazole capsule once in the morning before breakfast together with 3 tables of 2 mgs of Circadin (melatonin). In the evening, before dinner, patients will take 3 tablets of 2 mg of Circadin.
  Other Names: Circadin
  Arms: Melatonin + omeprazole

SUMMARY:
The study consists on determining whether melatonin decreases oxidative stress in Barrett's esophageal mucosa after 6 months of treatment. In order to achieve the clinical trial, the patients will be randomized to two possible arms: omeprazole alone or omeprazole plus melatonin. The patients will be followed around four visits during six months.

GERD is one of the most prevalent pathologies in the digestive tract. Barrett's esophagus, a complication of chronic GERD, has attracted the attention of researchers due to its condition of pre-neoplastic lesion. At present, treatment of Barrett's patients is limited to acid inhibition with PPIs. Although there are several studies which indicate that treatment with PPIs could decrease the incidence of high grade dysplasia and EAC, treatment with PPIs does not eliminate the risk of EAC in these patients. Therefore, it is necessary to find chemo-preventive agents that stop neoplastic progression of Barrett's esophagus. Among them, antioxidants have become the most promising agent. This pilot study will determine the efficacy of melatonin in the chemoprevention of EAC.

So, the main objective of this study is to determine whether melatonin decreases oxidative stress in Barrett's esophageal mucosa after 6 months of treatment.

To evaluate whether melatonin modifies other mechanisms associated to neoplastic progression in BE patients: proliferation and apoptotic index and molecular markers of progression: 17pLOH, 9pLOH, p16 methylation and DNA ploidy (tetraploidy and/or aneuploidy).

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a chronic disease secondary to the presence of stomach acid into the esophagus. This atypical situation produces an inflammation and ulceration of the distal esophagus mucosa. It is the main factor predisposing to the development of esophageal adenocarcinoma, which has a very poor prognosis. At present, therapy of Barrett's esophagus is based on acid secretion inhibition with proton pump inhibitors, which is a very effective therapy to reduce gastroesophageal reflux. However, this therapy does not completely eliminate this risk. Therefore, the better way to follow this disorder is to perform periodic upper gastrointestinal endoscopy and biopsies. Therefore, it is necessary to find new chemo-preventive agents that avoid more efficiently the neoplastic progression of BE. New advances in knowledge about BE suggest that antioxidants could be used to reduce the disorder development. These drugs are being used for long time ago in different pathologies in a lot of countries. One of these drugs is melatonin, which combines several characteristics that suggest it could be the most suitable antioxidant. It has no adverse effects reported.

Patients that meet the following characteristics will be included in this clinical study: Patients (males and females) with Barrett's esophagus (>18 years and <80) without macroscopic esophagitis at endoscopy and a length of the metaplasic mucosa of 2 cm or longer. By the same way, patients will be excluded of the study if present carcinoma or high grade dysplasia at basal endoscopy, previous gastric or esophageal surgery, patients on NSAID or aspirin treatment, neoplastic malignancies, hematological serious diseases (coagulation disorders and anemia with Hb < 9.5 gr/dL), serious/moderate cardiac, liver or renal diseases, need of corticosteroid therapy (a minimum of 5 days per month is allowed, as well as topical or inhaled treatment), patients on misoprostol or anticoagulants, patients with inflammatory bowel disease and allergy to investigational drugs.

Patients, who agree to participate in the study and meet criteria, will be randomized to one of the two following therapies: omeprazole alone or omeprazole + Circadin (melatonin.).

This intervention hardly produces any adverse effects, the most frequent adverse effects of proton pump inhibitors are headache and stomach ache. For melatonin has not reported any adverse effect.

This study will be done in the Hospital Clinico Lozano Blesa (Zaragoza, Spain), promoted by the Health Science Aragon Institute and its principal investigator is Angel Lanas Arbeloa (Digestive Disease Service). It will start in March-april 2012 and will finish 12 months later approximately. The study sponsor is I+CS (Aragon Institute of Health Sciences) that carries the cost of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients (males and females) with Barrett's esophagus (>18 years and <80) without macroscopic esophagitis at endoscopy and a length of the metaplasic mucosa of 2 cm or longer, who agree to participate in the study.

Exclusion Criteria:

* Presence of carcinoma or high grade dysplasia at basal endoscopy.
* Previous gastric or esophageal surgery.
* Patients on NSAID or aspirin treatment. A maximum of 5 days per month is allowed. Paracetamol will be used as the standard analgesic treatment.
* Neoplastic malignancies.
* Hematological serious diseases. Coagulation disorders and anemia with Hb < 9.5 gr/dL.
* Serious/moderate cardiac, liver or renal diseases.
* Need of corticosteroid therapy. A minimum of 5 days per month is allowed, as well as topical or inhaled treatment.
* Patients on misoprostol or anticoagulants.
* Patients with inflammatory bowel disease.
* Allergy to investigational drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | 6 months
  1. Peroxynitrite production. This variable will be measured by IHQ with a monoclonal Ab against nitrotyrosine residues in biopsy specimens taken from the metaplastic mucosa of patients with Barrett's esophagus.
  2. DNA oxidative damage: We will determine levels of 8-hydroxy-2'-deoxyguanosine in biopsy specimens form patients with Barrett's esophagus, as described above. DNA will be extracted with a commercial kit from Qiagen. 8-hydroxy-2'-deoxyguanosina quantification will be carried out by EIA.

SECONDARY OUTCOMES:
Biological markers of diseases progression | 6 months
  1. Cell proliferation (Ag ki67-mib1) measured by automatic morphometry NIH-Image 6.1).
  2. Apoptosis: measured by IHQ with caspase.
  3. Molecular markers of neoplastic progression.
The presence of DNA anomalies (tetraploidy and aneuploidy. | 6 months
  It will be determined by static cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Lanas Arbeloa, Physician, Principal Investigator — Digestive disease service of Hospital Clinico Lozano Blesa
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Spain